CLINICAL TRIAL: NCT05867147
Title: A Phase 1, Randomized, Double-blind, Placebo- and Positive-controlled, Thorough QT/QTc Study of Vanzacaftor Monotherapy in Healthy Subjects
Brief Title: An Electrocardiogram Study to Evaluate the Effect of Vanzacaftor on the QT/QTc Interval in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VX22-121-013
Record Dates: First submitted 2023-04-21; First posted 2023-05-19 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — deutivacaftor, tezacaftor , vanzacaftor; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Participants will receive VNZ-matching placebo, moxifloxacin-matching placebo and VNZ at different time points.
  Interventions: Drug: Vanzacaftor; Drug: Vanzacaftor Placebo; Drug: Moxifloxacin Placebo
- Group 2A (Active Comparator): Participants will receive VNZ-matching placebo, moxifloxacin, and moxifloxacin-matching placebo at different time points.
  Interventions: Drug: Vanzacaftor Placebo; Drug: Moxifloxacin; Drug: Moxifloxacin Placebo
- Group 2B (Active Comparator): Participants will receive VNZ-matching placebo, moxifloxacin-matching placebo and moxifloxacin at different time points.
  Interventions: Drug: Vanzacaftor Placebo; Drug: Moxifloxacin; Drug: Moxifloxacin Placebo

INTERVENTIONS:
Drug: Vanzacaftor — Tablets for oral administration.
  Arms: Group 1
Drug: Vanzacaftor Placebo — Placebo for oral administration.
Drug: Moxifloxacin — Tablets for oral administration.
  Arms: Group 2A; Group 2B
Drug: Moxifloxacin Placebo — Tablets for oral administration.

SUMMARY:
The purpose of this study is to evaluate the effect of Vanzacaftor (VNZ) on QTcF, as well as the pharmacokinetic (PK), safety, and tolerability of VNZ in healthy participants.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) of 18.0 to 32.0 kilogram per meter square (Kg/m^2), both inclusive
* Male and female participants of age 18 to 45 years, both inclusive
* Serum potassium, calcium, and magnesium values within normal ranges

Key Exclusion Criteria:

* Median QTcF>450 msec on triplicate 12-lead ECGs
* History of conduction abnormalities

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-06-14 (Actual)

PRIMARY OUTCOMES:
Change in QT interval corrected by Fridericia's formula (QTcF) | From Baseline up to Day 23

SECONDARY OUTCOMES:
Change in Heart Rate (HR) | From Baseline up to Day 23
Change in PR interval, segment | From Baseline up to Day 23
Change in QRS duration | From Baseline up to Day 23
Placebo-corrected Change in QTcF | From Baseline up to Day 23
Placebo-corrected Change in HR | From Baseline up to Day 23
Placebo-corrected Change in PR interval | From Baseline up to Day 23
Placebo-corrected Change in QRS duration | From Baseline up to Day 23
Number of Outliers for QTcF | From Baseline up to Day 23
Number of Outliers for HR | From Baseline up to Day 23
Number of Outliers for PR interval | From Baseline up to Day 23
Number of Outliers for QRS duration | From Baseline up to Day 23
Frequency of Treatment-emergent Changes of T-wave Morphology and U-wave Presence | From Baseline up to Day 23
Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day -2 up to Day 38
Maximum Observed Plasma Concentration (Cmax) of VNZ | Days 11 and 21
Area Under the Concentration Versus Time Curve From the Time of Dosing Extrapolated to 24 hours (AUC0-24h)) of VNZ | Days 11 and 21
Time Taken for VNZ to Reach Maximum Concentration (tmax) | Days 11 and 21

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion - Tempe, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing